CLINICAL TRIAL: NCT04733014
Title: Perceptions of Greek Ophthalmologists Regarding Contemporary Presbyopia Management.
Brief Title: Perceptions of Ophthalmologists Regarding Contemporary Presbyopia Management.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor, Democritus University of Thrace
Other Study IDs: ES1/Th3/21-1-2021
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Presbyopia
Keywords: Presbyopia, disease management, ophthalmologist, attitudes
MeSH Terms: conditions — Presbyopia; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Different attitudes and perceptions are encountered concerning contemporary presbyopia management. Exploration of ophthalmologists' attitudes on diagnostic and therapeutic management of presbyopia is essential for the development of disease management interventions by the Hellenic Ministry of Health and Welfare. Within this context, Greek ophthalmologists' perceptions on presbyopia will be explored by means of a custom questionnaire.

DETAILED DESCRIPTION:
Different attitudes and perceptions are encountered concerning contemporary presbyopia management. Exploration of ophthalmologists' attitudes on diagnostic and therapeutic management of presbyopia is essential for the development of disease management interventions by the Hellenic Ministry of Health and Welfare. Within this context, Greek ophthalmologists' perceptions on presbyopia will be explored by means of a custom questionnaire (DePrePer31).

ELIGIBILITY:
Inclusion Criteria:

* Valid license to practice ophthalmology in European Union.
* Adequate literacy of Greek language.

Exclusion Criteria:

* Pediatric ophthalmologist.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study's sample will be representative in terms of age, gender, geographic location.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-02-07 (Estimated); Study Completion 2021-02-07 (Estimated)

PRIMARY OUTCOMES:
Perceptions on presbyopia | 1 month
  Greek ophthalmologists' attitudes on contemporary presbyopia management

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, Study Chair — Democritus University of Thrace
Locations (1):
- Democritus University of Thrace, Alexandroupoli, Evros, Greece